CLINICAL TRIAL: NCT02206477
Title: DMSO for Prevention of Capsular Contraction in Alloplastic Breast Reconstruction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Sagit Meshulam-Derazon, MD; Head of breast reconstruction unit, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0005-13-RMC
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Breast Capsular Contracture; Dimethyl Sulfoxide
Keywords: breast capsular contructure; dimethyl sulfoxide; radiotherapy; breast reconstruction
MeSH Terms: interventions — Dimethyl Sulfoxide; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DMSO treatment group (Experimental): The treatment group will be exposed to DMSO according to our built protocol. On the seventh post-operative day, the patient will be guided to set 10 cc of DMSO soaked gauze compresses on the breast, twice a day for 20 minutes, for the term of 6 weeks. This treatment will be holed for 24 hours on tissue expander inflation dates. A repeated course of compresses will be taken after adjuvant radiotherapy, starting 24 hours after the last therapy.
  Interventions: Drug: Dimethyl Sulfoxide
- the control group (Placebo Comparator): The control group will be treated with the same post-operative protocol, but with 0.9% saline instead of DMSO. On the seventh post-operative day, the patient will be guided to set 10 cc 0.9% saline soaked gauze compresses on the breast, twice a day for 20 minutes, for the term of 6 weeks. This treatment will be holed for 24 hours on tissue expander inflation dates. A repeated course of compresses will be taken after adjuvant radiotherapy, starting 24 hours after the last therapy.
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Dimethyl Sulfoxide
  Other Names: DMSO
  Arms: DMSO treatment group
Drug: Saline 0.9%
  Other Names: normal saline
  Arms: the control group

SUMMARY:
Capsular contraction is the one of the most common complications of both esthetic and reconstructive breast surgery, with high incidence after radiotherapy. The mechanism of the contraction is unclear, but is believed to be similar to the formation of hypertrophic scarring.

Dimethyl sulfoxide (DMSO) has demonstrated its use as an anti-inflammatory, anti-proliferative, and antibacterial agent.

The aim of this study is to test the effect of DMSO on the incidence and severity if capsular contracture after breast alloplastic reconstruction in irradiated patients.

We conduct a prospective randomized-control single-surgeon study in the tertiary academic Rabin Medical Center.

110 female candidates for mastectomy, radiotherapy and immediate two-stage reconstruction will be included. They will be divided into two groups: the DMSO treatment group, which will be treated according to our protocol, and the control group, that will be treated with the same protocol but with 0.9% saline instead.

Several measures will be taken, including: capsular contracture grading by two plastic surgeons, a VAS-score of breast pain, maximal capsular thickness (MCT) in sonography evaluation, and pathology examination of the capsule (biopsy will be taken during the second stage operation).

Rates and grades of capsular contracture evident clinically, radiologically and pathologically, will be evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* female candidates for mastectomy, radiotherapy and immediate two-stage reconstruction

Exclusion Criteria:

* autologous reconstruction
* single-stage alloplastic reconstruction
* intake of steroids, anti-inflammatory, anti-coagulate or immunomodulatory medications on a regular basis
* low compliance to home treatment or follow-ups.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
reduction of 50% or more in capsular contructure incidence | 3.5 years

SECONDARY OUTCOMES:
reduction in maximal capsular thickness (MCT) in sonography evaluation | 3.5 years
evidence of less inflamation and fibrosis in pathology examination of the capsule | 3.5 years
reduction in VAS pain score in treatment group | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sagit Meshulam Derazon, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel